CLINICAL TRIAL: NCT03676166
Title: Pharmacokinetic and Pharmacodynamic Effects of Smoked and Vaporized Cannabis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB_00035394
Record Dates: First submitted 2018-09-16; First posted 2018-09-18 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-09

CONDITIONS: Cannabis
Keywords: Cannabis; Toxicology; Intoxication
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 0mg THC smoked cannabis (Experimental): placebo smoked cannabis
  Interventions: Drug: Cannabis
- 10mg THC smoked cannabis (Experimental): smoked cannabis containing 10mg THC
  Interventions: Drug: Cannabis
- 25mg THC smoked cannabis (Experimental): smoked cannabis containing 25mg THC
  Interventions: Drug: Cannabis
- 0mg THC vaporized cannabis (Experimental): placebo vaporized cannabis
  Interventions: Drug: Cannabis
- 10mg THC vaporized cannabis (Experimental): vaporized cannabis containing 10mg THC
  Interventions: Drug: Cannabis
- 25mg THC vaporized cannabis (Experimental): vaporized cannabis containing 25mg THC
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Cannabis — Inhaled cannabis

SUMMARY:
Few studies have been conducted to assess the pharmacokinetic and pharmacodynamic effects of smoked and vaporized cannabis. Careful analysis of different cannabis administration methods on these parameters is required to determine the level and duration of biological cannabinoid exposure and associated subjective, cardiovascular and cognitive effects. In the present study the investigators evaluated the detection of cannabinoids in whole blood, oral fluid, and urine, as well as the acute pharmacodynamics associated with smoked and vaporized cannabis among individuals who were not regular cannabis users. The outcomes of the study will extend scientific knowledge about the behavioral pharmacology and toxicology of smoked and vaporized cannabis administration and can inform policies regarding clinical, workplace and roadside drug testing programs.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written informed consent
2. Be between the ages of 18 and 45
3. Be in good general health based on a physical examination, medical history, vital signs, 12-lead ECG and screening urine and blood tests
4. Test negative for recent cannabis use in urine at the screening visit (confirmed by GC/MS laboratory test) and at clinic admission
5. Test negative for other drugs of abuse, including alcohol at the screening visit and at clinic admission
6. Not be pregnant or nursing (if female). All females must have a negative serum pregnancy test at the screening visit and a negative urine pregnancy test at clinic admission.
7. Have a body mass index (BMI) in the range of 19 to 36 kg/m2
8. Blood pressure at Screening Visit does not exceed a systolic blood pressure (SBP) of 150 mmHg or a diastolic blood pressure (DBP) of 90 mmHg

Exclusion Criteria:

1. Non-medical use of psychoactive drugs other than, nicotine, alcohol, or caffeine 3 month prior to the Screening Visit;
2. History of or current evidence of significant medical or psychiatric illness judged by the investigator to put the participant at greater risk of experiencing an adverse event due to exposure or completion of other study procedures.
3. Use of an OTC, systemic or topical drug(s), herbal supplement(s), or vitamin(s) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
4. Use of a prescription medication (with the exception of birth control prescriptions) within 14 days of experimental sessions; which, in the opinion of the investigator or sponsor, will interfere with the study result or the safety of the subject.
5. Use of hemp seeds or hemp oil in any form in the past 3 months.
6. Use of dronabinol (Marinol) within the past 6 months.
7. History of xerostomia (dry mouth), or the presence of mucositis, gum infection or bleeding, or other significant oral cavity disease or disorder that in the investigator's opinion may affect the collection of oral fluid samples.
8. History of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina).
9. Abnormal EKG result that in the investigator's opinion is clinically significant.
10. Enrolled in another clinical trial or have received any drug as part of a research study within 30 days prior to dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06-16 (Actual); Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Quantity of THC in blood | 8 hours post exposure
  Quantitative measurement of blood THC by LC-MS/MS

SECONDARY OUTCOMES:
Subjective rating of "Drug Effect" | 8 hours post exposure
  Visual Analog Scale rating of subjective drug effect. Score ranges from 0 (none) to 100 (extreme) using a 100mm line anchored with none/extreme designation.
Psychomotor performance as assessed by Digit Symbol Substitution Task | 8 hours post exposure
  Computerized version of Digit Symbol Substitution Task administered, total correct trials in 90-seconds measured
Memory performance as assessed by Paced Auditory Serial Addition Task | 8 hours post exposure
  Computerized version of Paced Auditory Serial Addition Task administered, total correct trials out of 90 recorded
Performance on Divided Attention Task | 8 hours post exposure
  Computerized Divided Attention Task administered, mean distance from central stimulus and number of targets correct out of 24 recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, PhD, Principal Investigator — Johns Hopkins School of Medicine Behavioral Pharmacology Research Unit
Locations (1):
- Johns Hopkins School of Medicine Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Spindle TR, Cone EJ, Schlienz NJ, Mitchell JM, Bigelow GE, Flegel R, Hayes E, Vandrey R. Acute Effects of Smoked and Vaporized Cannabis in Healthy Adults Who Infrequently Use Cannabis: A Crossover Trial. JAMA Netw Open. 2018 Nov 2;1(7):e184841. doi: 10.1001/jamanetworkopen.2018.4841. PMID 30646391